CLINICAL TRIAL: NCT00776295
Title: Phase II Trial of Autologous Peripheral Blood Hematopoietic Cell Transplantation (PBHCT) Followed by Dendritic Cell p53 Vaccination and Adoptive T Cell Transfer in Patients With Limited Stage Small Cell Lung Cancer
Brief Title: Autologous SCT Followed by Dendritic Cell p53 Vaccination in Patients With Limited Stage Small Cell Lung Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Low accrual
Sponsor: H. Lee Moffitt Cancer Center and Research Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MCC 14955; NCT00609583 (obsolete NCT alias)
Record Dates: First submitted 2008-10-20; First posted 2008-10-21 (Estimated); Results first posted 2012-06-21 (Estimated); Last update posted 2013-01-24 (Estimated); Status verified 2013-01

CONDITIONS: Small Cell Lung Cancer
Keywords: Small Cell Lung Cancer; SCLC; Limited Stage Small Cell Lung Cancer
MeSH Terms: conditions — Small Cell Lung Carcinoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- adeno virus vectored p53 (Experimental): Combined adenovirus vectored p53 tranfected dedritic cell vaccine and ex vivo expanded T-lymphocytes
  Interventions: Biological: Combined adenovirus vectored p53 tranfected dedritic cell vaccine and ex vivo expanded T-lymphocytes

INTERVENTIONS:
Biological: Combined adenovirus vectored p53 tranfected dedritic cell vaccine and ex vivo expanded T-lymphocytes — Autologous Dendritic Cells Derived from Peripheral Blood Mononuclear Cells, Cultured with Granulocyte-Macrophage Colony-Stimulating Factor and Interleukin 4, Transfected with Adenovirus Vector (Ad5CMV-p53, Introgen Therapeutics) Expressing Wildtype p53 Gene; Combined with Autologous Expanded T Lymphocytes (CD3+, CD4+, and CD8+), Cultured with OKT3 (Orthoclone) and Anti-CD28 (Repligen) Coated Magnetic Beads

SUMMARY:
The purpose of this study is to determine whether p53 vaccination followed by high dose chemotherapy and autologous HCT and T cell therapy significantly induces immune responses resulting in 1-year survival greater that the current 70%.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed SCLC who presented with Limited Stage (LS) at diagnosis.
* Measurable disease at the time of initial therapy
* Appropriate treatment for LS-SCLC including radiotherapy and chemotherapy.
* Responsive disease to standard chemoradiation therapy as defined by RECIST
* Patients with CR after chemoradiation therapy are strongly recommended to be treated with prophylactic cranial irradiation
* CBC with an absolute neutrophil count (ANC) >/= 1,000/uL, hemoglobin >/= 8.0 g/DL and platelet count >/= 75,000/uL.
* Normal prothrombin time (PT) and partial thromboplastin time (aPTT), unless on monitored anticoagulation therapy for medical conditions not excluded in the trial.
* Liver enzymes: total bilirubin less than or equal to 2mg/dL; AST and ALT less than 1.5X the upper limit of normal.
* Creatinine clearance of >/= 60 mL/min
* Pulmonary: DLCO greater than 50%
* Cardiac: left ventricular ejection fraction greater than 45%

Exclusion Criteria:

* Patient with stable (SD) or progressive disease (PD) after 4 cycles of standard cisplatin and etoposide and concurrent chest irradiation
* Pregnant or lactating woman
* HIV infection confirmed by NAT
* Common variable immunodeficiency
* Active CNS malignancy
* Active bacterial, fungal or viral infection
* Unfavorable psychosocial evaluation or history of poor compliance to prescribed medical care
* Prior history of autologous or allogeneic hematopoietic cell transplantation
* Presence of protocol specific comorbid conditions

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2007-05; Primary Completion 2010-06 (Actual); Study Completion 2010-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed Kharfan-Dabaja, MD, Principal Investigator — H. Lee Moffitt Cancer Center
Locations (1):
- HLeeMoffitt, Tampa, Florida, United States

REFERENCES:
- See also: H. Lee Moffitt Cancer Center & Research Institute — http://www.moffitt.org/

RESULTS

PARTICIPANT FLOW:
Groups:
- p53 Vaccination: Dendritic cell p53 vaccination
Period: Overall Study
Arm/Group | p53 Vaccination
Started | 2
Completed | 2
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | p53 Vaccination
Number analyzed (Participants) | 2
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 2
  >=65 years | 0
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 2
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 1
Region of Enrollment [Number; unit: participants]
  United States | 2

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects Meeting 1-year Overall Survival
Description: Number of participants with overall survival from first day of cyclophosphamide and GM-CSF mobilization to the day of death
Time Frame: up to one year
Measure: Number; unit: participants
Arm/Group | p53 Vaccination
Number analyzed (Participants) | 2
participants | 2

2. Secondary Outcome: 3 Year Progression-free Survival
Description: 3 year progression-free survival (PFS) is defined as time from maximum response to relapse or progression of SCLC
Time Frame: up to 3 years
Measure: Number; unit: participants
Arm/Group | p53 Vaccination
Number analyzed (Participants) | 2
participants | 0

ADVERSE EVENTS:
Groups:
- Biological/Vaccine: Combined adenovirus vectored p53 tranfected dedritic cell vaccine and ex vivo expaned T-lymphocytes
Arm/Group | Biological/Vaccine
Serious Adverse Events (participants affected / at risk) | 0/2
Other Adverse Events (participants affected / at risk) | 0/2

LIMITATIONS AND CAVEATS:
Early termination of trial due to small number of subjects thus leading to unreliabe data

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No